CLINICAL TRIAL: NCT03539185
Title: Airtraq Versus Fiberoptic for Awake Tracheal Intubation : A Randomised Non-inferiority Trial
Brief Title: Airtraq Versus Fiberoptic for Awake Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A00239-46
Record Dates: First submitted 2018-05-12; First posted 2018-05-29 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-05

CONDITIONS: Intubation;Difficult; Awake Intubation; Airway Complication of Anesthesia
Keywords: Airtraq; Fiberoptic; Awake; Tracheal intubation; laryngeal nerve blocks; sedation; remifentanil

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial. Alpha risk de 2,5%, Power 90 %
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airtraq (Active Comparator): Awake tracheal intubation using airtraq videolaryngoscope.
  Interventions: Device: Videolaryngoscope Airtraq
- Fiberoptic (Active Comparator): Awake nasotracheal tracheal intubation using flexible fiberoptic bronchoscope.
  Interventions: Device: Fiberoptic bronchoscope

INTERVENTIONS:
Device: Videolaryngoscope Airtraq — Awake orotracheal intubation with laryngeal nerve block and remifentanil sedation
  Arms: Airtraq
Device: Fiberoptic bronchoscope — Awake nasotracheal intubation with laryngeal nerve block and remifentanil sedation
  Arms: Fiberoptic

SUMMARY:
The airway management is a vital act in anesthesia. The gold standard technique for planned very difficult intubation is nasotracheal fiberoptic intubation. The success rate with this procedure is 98.8%. However, learning this technique is difficult and it's considered uncomfortable by patients and practitioners.

The Airtraq® videolaryngoscope is commonly used for difficult orotracheal intubation. Cases of awake intubation by Airtraq® have been described.

Furthermore, the French Society of Anesthesia-Resuscitation, in its last formalized expert recommendations (2017) on difficult intubation, proposes the use of video laryngoscopes as an alternative to the fiberoptic bronchoscope.

We propose a non-inferiority study evaluating the use of Airtraq® for the realization of a awake intubation compared to the gold standard (fiberoptic bronchoscope). This prospective randomized study should include 78 patients in two groups. The purpose of this study is to improve the comfort of patient and practitioner during an awake tracheal intubation, to facilitate the learning of the technique.

ELIGIBILITY:
Inclusion Criteria:

* Formal indication of awake intubation or patient with two criteria of difficult intubation and ventilation
* Major patient
* Patient able to understand oral and written information

Exclusion Criteria:

* Mouth opening (inter-incisor distance) <16 mm does not allow insertion of the Airtraq® videolaryngoscope
* Surgery requires nasotracheal intubation
* Loco-regional anesthesia of larynx impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Success of orotracheal or nasotracheal intubation. | 1 day
  Defined by the visualization of the tube into the trachea through vocal cords and by the appearance of the capnogram

SECONDARY OUTCOMES:
Length of the proceedings | 1 day
  Duration between the insertion of device and the appearance of capnogram
Rate of occurrence of adverse events | 1 day
  Coughing, desaturation, agitation
Patient satisfaction score | 1 day
  Analogue visual scale graduated from zero to ten. Zero is the worst imaginable satisfaction and 10 is the better imaginable satisfaction.
Operator satisfaction score | 1 day
  Analogue visual scale graduated from zero to ten. Zero is the worst imaginable satisfaction and 10 is the better imaginable satisfaction.
Number of intubation attempts | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre FRUGIER, Résident, Principal Investigator — University Hospital, Caen; Hervé KAMGA, Dr, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU de Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Collins SR, Blank RS. Fiberoptic intubation: an overview and update. Respir Care. 2014 Jun;59(6):865-78; discussion 878-80. doi: 10.4187/respcare.03012. PMID 24891196
- [Result] Pintaric TS. UPPER AIRWAY BLOCKS FOR AWAKE DIFFICULT AIRWAY MANAGEMENT. Acta Clin Croat. 2016 Mar;55 Suppl 1:85-9. PMID 27276778
- [Result] Law JA, Morris IR, Brousseau PA, de la Ronde S, Milne AD. The incidence, success rate, and complications of awake tracheal intubation in 1,554 patients over 12 years: an historical cohort study. Can J Anaesth. 2015 Jul;62(7):736-44. doi: 10.1007/s12630-015-0387-y. Epub 2015 Apr 24. PMID 25907462
- [Result] Law JA, Morris IR, Milne AD. The complications of awake tracheal intubation. Can J Anaesth. 2015 Sep;62(9):1023. doi: 10.1007/s12630-015-0402-3. Epub 2015 May 12. No abstract available. PMID 25963612
- [Result] Allan AG. Reluctance of anaesthetists to perform awake intubation. Anaesthesia. 2004 Apr;59(4):413. doi: 10.1111/j.1365-2044.2004.03729.x. No abstract available. PMID 15023129
- [Result] Xu YC, Xue FS, Luo MP, Yang QY, Liao X, Liu Y, Zhang YM. Median effective dose of remifentanil for awake laryngoscopy and intubation. Chin Med J (Engl). 2009 Jul 5;122(13):1507-12. PMID 19719938
- [Result] Dawson AJ, Marsland C, Baker P, Anderson BJ. Fibreoptic intubation skills among anaesthetists in New Zealand. Anaesth Intensive Care. 2005 Dec;33(6):777-83. doi: 10.1177/0310057X0503300613. PMID 16398385
- [Result] Dimitriou VK, Zogogiannis ID, Liotiri DG. Awake tracheal intubation using the Airtraq laryngoscope: a case series. Acta Anaesthesiol Scand. 2009 Aug;53(7):964-7. doi: 10.1111/j.1399-6576.2009.02012.x. Epub 2009 Jun 3. PMID 19496763
- [Result] Suzuki A, Toyama Y, Iwasaki H, Henderson J. Airtraq for awake tracheal intubation. Anaesthesia. 2007 Jul;62(7):746-7. doi: 10.1111/j.1365-2044.2007.05155.x. No abstract available. PMID 17567358